CLINICAL TRIAL: NCT07206329
Title: A Prospective Study Comparing Ultra-Low Volume Bowel Preparations for Capsule Colonoscopy and Pan-Intestinal Capsule Endoscopy: Efficacy of 1L Polyethylene Glycol Plus Ascorbic Acid vs. Sodium Picosulfate With Magnesium Citrate
Brief Title: PEG-Asc Vs. SPMC for Bowel Preparation in Capsule-based Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde do Alto Ave, EPE (Other)
Responsible Party: Principal Investigator, João Carlos Lima Gonçalves, MDPhD, Unidade Local de Saúde do Alto Ave, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 64/2024
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bowel Preparation Solution
Keywords: Capsule Colonoscopy; Pan-intestinal Capsule Endoscopy; Bowel Cleansing; Ultra-low-volume Bowel Preparation; Polyethylene Glycol plus Ascorbic Acid; Sodium Picosulfate with Magnesium Citrate
MeSH Terms: interventions — Polyethylene Glycols; Ascorbic Acid; picosulfate sodium; magnesium citrate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyethylene Glycol plus Ascorbic Acid (PEG-Asc) (Experimental): Participants receive a split-dose bowel preparation with 1 L polyethylene glycol plus ascorbic acid (PEG-Asc). The first dose is administered at 20:00 the evening before the procedure (500 mL PEG-Asc solution consumed over 1 hour, followed by 500 mL clear liquids). The second identical dose is taken at 06:00 on the day of the capsule procedure.
  Interventions: Drug: Polyethylene Glycol plus Ascorbic Acid (PEG-Asc)
- Sodium Picosulfate with Magnesium Citrate (SPMC) (Experimental): Participants receive a split-dose bowel preparation with sodium picosulfate and magnesium citrate (SPMC). The first dose is administered at 20:00 the evening before the procedure (1 sachet dissolved in 150 mL water, followed by 1.5-2 L clear liquids over 1-2 hours). The second identical dose is taken at 06:00 on the day of the capsule procedure.
  Interventions: Drug: Sodium Picosulfate with Magnesium Citrate (SPMC)

INTERVENTIONS:
Drug: Polyethylene Glycol plus Ascorbic Acid (PEG-Asc) — Participants receive a split-dose bowel preparation with 1 L polyethylene glycol plus ascorbic acid (PEG-Asc). The first dose is administered at 20:00 the evening before the procedure (500 mL PEG-Asc solution consumed over 1 hour, followed by 500 mL clear liquids). The second identical dose is taken at 06:00 on the day of the capsule procedure.
  Other Names: 1L PEG with Ascorbate
  Arms: Polyethylene Glycol plus Ascorbic Acid (PEG-Asc)
Drug: Sodium Picosulfate with Magnesium Citrate (SPMC) — Participants receive sodium picosulfate with magnesium citrate (SPMC) in a split-dose regimen. The first sachet is dissolved in 150 mL water and followed by 1.5-2 L of clear fluids the evening before the procedure, and the second sachet is taken with the same fluid regimen on the morning of the procedure.
  Other Names: SPMC; Sodium Picosulfate + Mg Citrate
  Arms: Sodium Picosulfate with Magnesium Citrate (SPMC)

SUMMARY:
This clinical research study is designed to find out which of two different types of bowel preparation works best for people undergoing capsule-based endoscopy procedures. Capsule colonoscopy and pan-intestinal capsule endoscopy ("panendoscopy") are newer, less invasive tests that use a small camera inside a capsule that is swallowed, instead of a traditional colonoscopy that requires a long flexible tube. These tests allow doctors to see the inside of the colon, and in the case of panendoscopy, also the small intestine. They are especially useful when a regular colonoscopy cannot be completed or when doctors need to investigate conditions such as Crohn's disease, anemia, or unexplained bleeding.

For these capsule procedures to work well, the bowel needs to be as clean as possible, since the capsule cannot wash or suction away any stool or bubbles. This makes the type of bowel preparation very important, but at present there are no clear recommendations about which preparation to use. Standard preparations often involve large volumes of liquid that patients may find difficult to drink. In recent years, ultra-low-volume preparations (1 liter or less) have been developed to improve patient comfort and make the preparation process easier.

In this study, we are comparing two of these ultra-low-volume options: Polyethylene Glycol plus Ascorbic Acid (PEG-Asc), a 1-liter solution and Sodium Picosulfate with Magnesium Citrate (SPMC), a powder mixed with water.

We want to see which of these two preparations provides better bowel cleansing for capsule procedures, while also checking which is easier for patients to tolerate.

A total of 220 adult patients referred for capsule colonoscopy or panendoscopy were enrolled and randomly assigned to receive either PEG-Asc or SPMC. Both groups followed a split-dose schedule, with part of the preparation taken the evening before and part on the morning of the test, along with additional instructions including dietary restrictions, laxative tablets, and clear liquids.

The main questions this study is trying to answer are:

1. - Which preparation results in better cleaning of the bowel, allowing clearer pictures from the capsule?
2. - Which preparation is easier for patients to tolerate, with fewer side effects such as nausea or vomiting?
3. - Does the type of preparation affect whether the capsule can complete the examination and reach the end of the colon?

By answering these questions, this study hopes to improve the effectiveness and comfort of capsule endoscopy procedures. The results will help doctors decide which bowel preparation to recommend, making these less invasive tests more reliable and accessible for patients in the future.

DETAILED DESCRIPTION:
Capsule colonoscopy (CC) and pan-intestinal capsule endoscopy ("panendoscopy") are increasingly used diagnostic modalities in clinical practice. Capsule colonoscopy is most often indicated when a complete conventional colonoscopy cannot be achieved due to technical difficulties (looping, sharp angulation), patient intolerance, or contraindications to sedation. Panendoscopy allows simultaneous visualization of the small bowel and colon and is especially relevant in the diagnostic work-up of Crohn's disease and obscure gastrointestinal bleeding.

A key limitation of capsule-based procedures is the inability to wash or aspirate debris. Consequently, bowel preparation quality has a direct and critical impact on diagnostic yield. Residual stool, bubbles, or opaque fluid can obscure mucosal visualization, leading to missed lesions or inconclusive examinations. Meta-analyses of capsule endoscopy studies highlight substantial variability in preparation protocols, with pooled adequate cleansing rates around 70%. However, no standardized regimen has been established, and current practice often relies on multi-step protocols combining dietary restrictions, stimulant laxatives, split-dose purgatives, prokinetics, and booster solutions.

Traditional polyethylene glycol (PEG)-based regimens are effective but often require ingestion of large fluid volumes (2-4 liters), which reduces tolerability and adherence. Recently, ultra-low-volume regimens (≤1 L) have been developed, aiming to improve patient acceptance while maintaining cleansing efficacy. Among these, 1 L PEG plus ascorbic acid (PEG-Asc) and sodium picosulfate with magnesium citrate (SPMC) are widely used in conventional colonoscopy, where multiple randomized controlled trials and meta-analyses have shown them to be non-inferior to higher-volume preparations, with superior tolerability profiles. However, their performance in capsule-based procedures has not previously been tested.

The primary aim of this study was to compare the bowel cleansing efficacy of PEG-Asc and SPMC in patients undergoing capsule colonoscopy or panendoscopy. Secondary aims were to evaluate tolerability, adverse events, completion rates, and the prevalence of clinically relevant findings (polyps, diverticula, inflammatory changes, angioectasias).

This was a prospective, single-center, randomized, researcher-blinded clinical trial. Between January 2024 and June 2025, consecutive adult outpatients referred for CC or panendoscopy were enrolled and randomized in a 1:1 ratio to receive either PEG-Asc or SPMC. Randomization was performed using block allocation. Patients provided written informed consent prior to participation.

All patients discontinued iron supplementation one week before the procedure and followed a low-fiber diet two days before capsule ingestion. Oral senna 12 mg was administered twice daily for two days prior. After 2:00 PM on the day before the procedure, patients transitioned to a clear liquid diet.

PEG-Asc group: In the evening (8:00 PM), patients ingested 1 L solution consisting of 500 mL PEG-Asc taken over one hour, followed by 500 mL of clear fluids. The second dose was repeated at 6:00 AM on the day of the procedure.

SPMC group: In the evening, patients dissolved one sachet of SPMC in 150 mL water, ingested it, and followed with 1.5-2 L of clear fluids over 1-2 hours. The second sachet was taken at 6:00 AM in the same manner.

Patients received 10 mg domperidone 30 minutes before capsule ingestion. A PillCam™ COLON 2 or PillCam™ CROHN'S capsule was swallowed. Real-time viewer checks ensured small-bowel entry; if delayed, domperidone was repeated or endoscopic delivery was performed. Booster doses of sodium phosphate solution were administered to facilitate capsule propulsion (30 mL + 1 L water after small-bowel entry; 15 mL + 1 L water 3 hours later). Bisacodyl suppository was administered if the capsule had not been expelled after the scheduled meal.

Primary outcomes: Adequate bowel cleansing (assessed using the validated CC-CLEAR scale) and procedure completion rate (visualization of hemorrhoidal plexus or documented expulsion).

Secondary outcomes: Patient-reported tolerability (questionnaire), adverse events, compliance, and detection of clinically relevant findings (polyps, diverticula, inflammation, angioectasias).

Capsule videos were reviewed independently by two experienced readers blinded to allocation, using twin-head mode on RAPID® software. The colon was divided into right, transverse, and left segments, scored according to the percentage of mucosa visualized. Adequate cleansing was defined as all segments scoring ≥2 and an overall CC-CLEAR score ≥6. If any segment scored ≤1, the preparation was considered inadequate.

Continuous variables were tested for normality (Shapiro-Wilk). Normally distributed data were compared with Student's t-test; non-normal data with the Mann-Whitney U test. Categorical variables were analyzed using chi-square or Fisher's exact test. Significance was set at p<0.05 (two-tailed). Analyses were conducted using SPSS v28.

This trial addresses a critical gap in evidence regarding ultra-low-volume bowel preparation regimens for capsule endoscopy. Because capsule procedures cannot compensate for residual stool or fluid, optimal preparation is essential to ensure diagnostic accuracy and clinical utility. By comparing PEG-Asc and SPMC directly in this context, the study will provide much-needed data to inform best practices. Findings are expected to guide selection of bowel regimens in clinical practice, improve patient outcomes by optimizing mucosal visualization, and support the broader adoption of capsule-based diagnostics.

ELIGIBILITY:
Inclusion Criteria

* Adults referred for capsule colonoscopy (CC) or pan-intestinal capsule endoscopy (PCE)
* Ability to provide informed consent

Exclusion Criteria

* Contraindications to capsule endoscopy (e.g., known or suspected gastrointestinal obstruction, strictures, or fistulas)
* Contraindications to the use of PEG-Asc or SPMC (e.g., severe renal impairment, congestive heart failure, electrolyte disturbances, hypersensitivity to study drugs)
* Pregnancy or lactation
* Inability to comply with the bowel preparation protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Adequate bowel cleansing rate assessed by CC-CLEAR scale | Within 24 hours of capsule ingestion
  Proportion of patients achieving adequate overall bowel cleansing, defined as CC-CLEAR score ≥6 with no segment scoring ≤1.

SECONDARY OUTCOMES:
Capsule completion rate | Within 24 hours of capsule ingestion
  Proportion of procedures in which the capsule reached the hemorrhoidal plexus or was expelled during the recording period.
Patient tolerability | Day of procedure
  Patient-reported tolerability of bowel preparation using a 5-point scale ("very easy" to "very difficult").
Adverse events | Within 48 hours of capsule ingestion
  Frequency of adverse events including nausea, vomiting, headache, abdominal pain, or serious events requiring medical evaluation.
Detection of clinically relevant findings | Within 24 hours of capsule ingestion
  Proportion of patients with clinically relevant findings (polyps, diverticula, inflammation, or angioectasias) identified during capsule endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: José B Cotter, MD PhD, Study Director — Unidade Local de Saúde do Alto Ave
Locations (1):
- Unidade Local de Saúde do Alto Ave (ULSAAVE), Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this study will be made available upon reasonable request to the corresponding author. Access will be granted to researchers with methodologically sound proposals for use in scientific research, subject to approval and data-sharing agreements.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the primary manuscript and for a period of 5 years thereafter.
Access Criteria: Data will be shared through secure transfer after approval of a formal request submitted to the corresponding author.
URL: https://orcid.org/0000-0002-4081-8072

REFERENCES:
- [Background] Vuik FER, Nieuwenburg SAV, Moen S, Spada C, Senore C, Hassan C, Pennazio M, Rondonotti E, Pecere S, Kuipers EJ, Spaander MCW. Colon capsule endoscopy in colorectal cancer screening: a systematic review. Endoscopy. 2021 Aug;53(8):815-824. doi: 10.1055/a-1308-1297. Epub 2021 Jan 13. PMID 33440442
- [Background] Rosa B, Donato H, Curdia Goncalves T, Sousa-Pinto B, Cotter J. What Is the Optimal Bowel Preparation for Capsule Colonoscopy and Pan-intestinal Capsule Endoscopy? A Systematic Review and Meta-Analysis. Dig Dis Sci. 2023 Dec;68(12):4418-4431. doi: 10.1007/s10620-023-08133-7. Epub 2023 Oct 13. PMID 37833441